CLINICAL TRIAL: NCT05352243
Title: Combined Expressive Disclosure and Prosocial Writing to Promote Well-Being and Decrease Psychological Distress Among Bereaved Emerging Adults: Examining The Roles of Psychological Distancing, Universality, and Generativity
Brief Title: Bereaved Young Adults Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Brittany Drake, MA, CPhil, Principal Investigator, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 21-001728
Record Dates: First submitted 2022-04-22; First posted 2022-04-28 (Actual); Last update posted 2023-05-16 (Actual); Status verified 2023-05

CONDITIONS: Bereavement
Keywords: Expressive Disclosure; Prosocial; Expressive Writing; Peer Helping; Young Adults

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Expressive Disclosure (Active Comparator): Participants will be instructed to write about their deepest thoughts and feelings surrounding their bereavement experience.
  Interventions: Behavioral: Expressive Disclosure
- Expressive Helping (Experimental): Participants will be instructed to write about their deepest thoughts and feeling surrounding their bereavement experience in their first two essays and to provide advice and support for someone who recently experienced a loss in their final essay.
  Interventions: Behavioral: Expressive Helping
- Fact-Writing (Sham Comparator): Participants will be instructed to write objectively about different time frames (e.g., routine for getting up in the morning, routine for going to sleep at night).
  Interventions: Behavioral: Fact-Writing

INTERVENTIONS:
Behavioral: Expressive Disclosure — Prior to each writing session, participants will receive general instructions for completing the writing (e.g., write continuously for 20 minutes, do not worry about grammar, sentence structure, repetition), and be reminded that their writing will remain confidential. Three writing sessions will be spaced 1-2 weeks apart. A weekly writing prompt will instruct participants to write about their deepest thoughts and feelings surrounding their bereavement experience.
  Arms: Expressive Disclosure
Behavioral: Expressive Helping — Prior to each writing session, participants will receive general instructions for completing the writing (e.g., write continuously for 20 minutes, do not worry about grammar, sentence structure, repetition), and be reminded that their first two writing will remain confidential, and their final essay will be de-identified before being provided to newly bereaved young adults. Three writing sessions will be spaced 1-2 weeks apart. In the first two writing sessions, participants will receive a writing prompt that will instruct them to write about their deepest thoughts and feelings surrounding their bereavement experience. For the final writing session, participants will receive a writing prompt instructing them to provide advice and support for a newly bereaved young adult.
  Arms: Expressive Helping
Behavioral: Fact-Writing — Prior to each writing session, participants will receive general instructions for completing the writing (e.g., write continuously for 20 minutes, do not worry about grammar, sentence structure, repetition), and be reminded that their writing will remain confidential. Three writing sessions will be spaced 1-2 weeks apart. A weekly writing prompt will instruct participants to write objectively about different time frames (e.g., routine for getting up in the morning, routine for going to sleep at night).
  Arms: Fact-Writing

SUMMARY:
Bereaved adolescents and emerging adults are at risk for developing psychological disorders and complicated grief. Clinical grief interventions and conventional wisdom reflect an implicit assumption that sharing and expressing one's feelings surrounding a loss (i.e., emotional disclosure) facilitates psychological adjustment. However, studies of emotional disclosure have yielded null results in bereaved samples. Individuals who have encountered stressful life events, including interpersonal loss, often report a desire to "give back" to others in similar situations. Empirical evidence suggests that providing support to others can be equally, if not more, beneficial than receiving support. The opportunity to support others experiencing stressful circumstances may address common feelings of powerlessness and engender a sense of meaning, enhancing positive affect and reducing distress. Interventions that leverage prosocial behaviors are associated with positive effects, including increases in wellbeing in non-bereaved populations. To date, no research has examined the utility of prosocial interventions for bereaved individuals.

The present study tests a novel expressive helping intervention that combines elements of expressive disclosure and prosocial writing. Expressive helping will be compared to traditional expressive disclosure and a neutral writing control condition in a sample of bereaved young adults. Participants (N=156) will be randomized to one of three conditions-expressive disclosure, expressive helping, or a neutral writing control-and complete three weekly 20-minute writing sessions. Measures of psychological distress, well-being, and hypothesized mediators will be administered before, immediately following (within 48 hours of the final writing session), one month, and two months after the writing sessions. It is hypothesized that the participants in the expressive helping condition will evidence greater increases in well-being and decreases in grief-related distress at the one and two-month follow-ups, as compared to the other two groups.

ELIGIBILITY:
Inclusion Criteria:

1. Experienced the death of a loved one within the last 5 years, but more than 6 months ago.
2. Endorse having close relationship with loved one at time of their death (i.e., 5 or above on 1-10 likert scale with 1 being not at all close, and 10 being extremely close).
3. Endorse moderate to severe distress about the loss (i.e., 5 or above on 1-10 likert scale with 1 being not at all distressed, and 10 being extremely distressed).
4. Feel comfortable writing in English (due to the linguistic nature of the writing sessions).
5. Have access to the Internet and a computer to complete the assessments and writing sessions.

Exclusion Criteria:

1. Express active psychosis or suicidal ideation, or any other circumstances that, in the opinion of the investigators, compromise participant safety.

Ages: 18 Years to 26 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 178 (Actual)
Dates: Start 2022-01-24 (Actual); Primary Completion 2022-09-01 (Actual); Study Completion 2022-09-01 (Actual)

PRIMARY OUTCOMES:
Change in Wellbeing | Baseline (≤2 weeks of starting the intervention), post-intervention survey (≤1 week after the final writing assignment), the 1-month follow-up, and 2-month follow up.
  Wellbeing within the past two weeks will be measured at baseline, post-intervention, and the 1-month follow-up via the 14-item Mental Health Continuum-Short Form (MHC-SF; Keyes, 2009). The MHC-SF is comprised of three empirically derived subscales: the 3-item Emotional Well-Being Subscale, the 6-item Psychological Well-Being Subscale, and the 5-item Social Well-Being Subscale. Higher scores on each subscale, and the total score overall (range: 0-56), indicate greater well-being.
Change in Grief Reactions | Baseline (≤2 weeks of starting the intervention), post-intervention survey (≤1 week after the final writing assignment), the 1-month follow-up, and 2-month follow up.
  Grief-related distress within the past two weeks will be measured using the 18-item Traumatic-Grief Inventory Self-Report version (TGI-SR; Boelen et al., 2019). The TGI-SR includes items that reflect the criteria for Prolonged Grief Disorder (PGD) and Persistent Complex Bereavement Disorder set forth by the Diagnostic and Statistical Manual of Mental Disorders and International Classification of Diseases, respectively. Higher scores (range: 18-90) indicate more severe potentially impairing grief reactions.

SECONDARY OUTCOMES:
Change in Physical Symptoms | Baseline (≤2 weeks of starting the intervention), post-intervention survey (≤1 week after the final writing assignment), the 1-month follow-up, and 2-month follow up.
  Physical symptoms within the past two weeks will be measured using the Pennebaker Inventory of Limbic Languidness (PILL; Pennebaker et al., 1982). The PILL contains 54 items measured using a 5-point scale for the frequency of a variety of common physical symptoms (1 = never, 5 = more than once every week). Higher total scores (range, 0-216) indicate greater symptomatology.
Change in Anxiety | Baseline (≤2 weeks of starting the intervention), post-intervention survey (≤1 week after the final writing assignment), the 1-month follow-up, and 2-month follow up.
  Anxiety symptoms over the past 2 weeks will be measured using the 7-item PROMIS - Anxiety Short Form (Pilkonis, 2011). Higher scores (range: 7-35) on this scale indicate greater severity of anxiety symptoms.
Change in Depressive Symptoms | Baseline (≤2 weeks of starting the intervention), post-intervention survey (≤1 week after the final writing assignment), the 1-month follow-up, and 2-month follow up.
  Depressive symptoms over the past two weeks will be measured using the 20-item Center for Epidemiological Studies Depression Scale (CES-D; Radloff, 1977). The CES-D is a measure of symptom severity. Higher scores (range: 0-60) on this scale indicate greater depressive symptom severity.

OTHER OUTCOMES:
Change in Universality | Baseline (≤2 weeks of starting the intervention), directly after each writing session, post-intervention survey (≤1 week after the final writing assignment), the 1-month follow-up, and 2-month follow up.
  Feelings of universality over the past two weeks and during the writing sessions will be measured using adapted versions of items included in a questionnaire used in research regarding group therapy and social support groups (i.e., Weinberg et al., 1995, Yalom, 1995). Feelings of universality will be assessed with 3 items (e.g., "I feel understood and accepted by others who have experienced a loss."). A higher total score (range: 3-21) indicates greater feelings of universality.
Change in Psychological Distance | Baseline (≤2 weeks of starting the intervention), directly after each writing session, post-intervention survey (≤1 week after the final writing assignment), the 1-month follow-up, and 2-month follow up.
  Psychological distance while thinking and while completing the writing sessions will be measured using adapted items from previous research on psychological distance (i.e., Ayduk & Kross, 2010; Libby & Eibach, 2011; Ross & Wilson, 2002). Psychological will be assessed with 4 items. A higher total score (range: 4-28) indicates psychological distance.
Change in Generativity | Baseline (≤2 weeks of starting the intervention), directly after each writing session, post-intervention survey (≤1 week after the final writing assignment), the 1-month follow-up, and 2-month follow up.
  Feelings of generativity over the past two weeks and while completing the writing sessions will be measured using the 6-item generative achievement subscale of the Generativity Scale (Gruenewald et al., 2015). Higher scores (range: 13-78) on this scale indicate greater generativity levels.
Change in Coping Tendency | Baseline (≤2 weeks of starting the intervention), post-intervention survey (≤1 week after the final writing assignment), the 1-month follow-up, and 2-month follow up.
  Coping processes within the past two weeks will be measured using the COPE approach-oriented coping subscales (i.e., positive reinterpretation, emotional support, and acceptance; Carver et al., 1989), emotional approach coping scales (i.e., emotional processing, emotional expression; Stanton et al., 2000), and the COPE avoidance-oriented coping subscales (i.e., mental disengagement, denial; Carver et al., 1989; Eisenberg et al., 2012). Each subscale contains 4 times (28 items total) and assesses coping strategy use. Higher scores on each subscale (range: 4-16) indicate greater use of the associated coping strategy.

CONTACTS AND LOCATIONS:
Locations (1):
- University of California, Los Angeles, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ayduk O, Kross E. From a distance: implications of spontaneous self-distancing for adaptive self-reflection. J Pers Soc Psychol. 2010 May;98(5):809-29. doi: 10.1037/a0019205. PMID 20438226
- [Background] Boelen PA, Djelantik AAAMJ, de Keijser J, Lenferink LIM, Smid GE. Further validation of the Traumatic Grief Inventory-Self Report (TGI-SR): A measure of persistent complex bereavement disorder and prolonged grief disorder. Death Stud. 2019;43(6):351-364. doi: 10.1080/07481187.2018.1480546. Epub 2018 Jul 17. PMID 30015568
- [Background] Carver CS, Scheier MF, Weintraub JK. Assessing coping strategies: a theoretically based approach. J Pers Soc Psychol. 1989 Feb;56(2):267-83. doi: 10.1037//0022-3514.56.2.267. PMID 2926629
- [Background] Eisenberg SA, Shen BJ, Schwarz ER, Mallon S. Avoidant coping moderates the association between anxiety and patient-rated physical functioning in heart failure patients. J Behav Med. 2012 Jun;35(3):253-61. doi: 10.1007/s10865-011-9358-0. Epub 2011 Jun 10. PMID 21660588
- [Background] Gruenewald TL, Tanner EK, Fried LP, Carlson MC, Xue QL, Parisi JM, Rebok GW, Yarnell LM, Seeman TE. The Baltimore Experience Corps Trial: Enhancing Generativity via Intergenerational Activity Engagement in Later Life. J Gerontol B Psychol Sci Soc Sci. 2016 Jul;71(4):661-70. doi: 10.1093/geronb/gbv005. Epub 2015 Feb 25. PMID 25721053
- [Background] Keyes, C. L. M. (2009). Atlanta: Brief description of the mental health continuum short form (MHC-SF).
- [Background] Libby LK, Eibach RP. Looking back in time: self-concept change affects visual perspective in autobiographical memory. J Pers Soc Psychol. 2002 Feb;82(2):167-79. PMID 11831407
- [Background] Pennebaker JW, Gonder-Frederick L, Stewart H, Elfman L, Skelton JA. Physical symptoms associated with blood pressure. Psychophysiology. 1982 Mar;19(2):201-10. doi: 10.1111/j.1469-8986.1982.tb02547.x. No abstract available. PMID 7071299
- [Background] Pilkonis PA, Choi SW, Reise SP, Stover AM, Riley WT, Cella D; PROMIS Cooperative Group. Item banks for measuring emotional distress from the Patient-Reported Outcomes Measurement Information System (PROMIS(R)): depression, anxiety, and anger. Assessment. 2011 Sep;18(3):263-83. doi: 10.1177/1073191111411667. Epub 2011 Jun 21. PMID 21697139
- [Background] Radloff, L. S. (1977). The CES-D scale: A self-report depression scale for research in the general population. Applied psychological measurement, 1(3), 385-401.
- [Background] Ross M, Wilson AE. It feels like yesterday: self-esteem, valence of personal past experiences, and judgments of subjective distance. J Pers Soc Psychol. 2002 May;82(5):792-803. PMID 12003478
- [Background] Stanton AL, Kirk SB, Cameron CL, Danoff-Burg S. Coping through emotional approach: scale construction and validation. J Pers Soc Psychol. 2000 Jun;78(6):1150-69. doi: 10.1037//0022-3514.78.6.1150. PMID 10870915
- [Background] Weinberg, N., Uken, J. S., Schmale, J., & Adamek, M. (1995). Therapeutic factors: Their presence in a computer-mediated support group. Social Work with Groups, 18, 57-69.
- [Background] Yalom, I. D. (1995). The theory and practice of group psychotherapy. Basic Books.